CLINICAL TRIAL: NCT06560385
Title: A Pilot, Double-blind, Randomised, Placebo-controlled Trial on the Efficacy of a Synbiotic Formula (BLHK03) in Alleviating Chemotherapy-induced Alopecia (CIA) in Breast Cancer Patients
Brief Title: Alleviation of Alopecia in Breast Cancer Patient Using Synbiotics Formula
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GenieBiome Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BCIA Study
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Hair Loss
Keywords: Breast Cancer; Hair Loss; Chemotherapy; Synbiotic
MeSH Terms: conditions — Breast Neoplasms; Alopecia

STUDY DESIGN:
Intervention Model Description: All subjects will be randomized into two group to take BLHK03 or active placebo (Vitamin B7) daily from the start of the chemotherapy cycle to 2 months after the final dose of chemotherapy.
Who Masked: Participant, Investigator
Masking Description: Attending physicians, investigators performing assessments in clinic visits and study participants will be blinded to the group allocation until study completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Active Comparator): Subjects will receive 1 sachet of BLHK03 daily from the start of the chemotherapy cycle to 2 months after the final dose of chemotherapy.
  Interventions: Dietary Supplement: BLHK03
- Placebo arm (Placebo Comparator): Subjects will receive 1 sachet of active placebo daily from the start of the chemotherapy cycle to 2 months after the final dose of chemotherapy.
  Interventions: Dietary Supplement: Active placebo

INTERVENTIONS:
Dietary Supplement: BLHK03 — BLHK03 consists of a blend of probiotics (20 billion CFU in 1 sachet) and prebiotic compounds
  Arms: Active arm
Dietary Supplement: Active placebo — Active placebo contains 5mcg of Vitamin B7
  Arms: Placebo arm

SUMMARY:
This study aims to explore the efficacy and safety of a synbiotic formula (BLHK03) in alleviating chemotherapy-induced alopecia (CIA) in breast cancer patients and the compositional and functional changes in the gut microbiome of breast cancer patients undergoing chemotherapy and treatment with BLHK03.

DETAILED DESCRIPTION:
In a mice study, it was shown that oral administration of a probiotic isolated from healthy faeces, B. longum HK003, has protective effects against alopecia related to chemotherapy. Mice were treated with 100 mg/kg cyclophosphamide (CYP) once monthly, for 4 months. The CYP-treated mice were then treated with B. longum HK003 for 14 days. Results showed that B. longum treatment significantly enhanced skin thickness histologically. In the subcutis, the quantity and size of anagen follicles were increased, whilst the quantity of atrophic follicles were decreased.

Currently, there is no documentation of potential probiotic-drug interactions in breast cancer patients undergoing chemotherapy. A previous randomized controlled trial reported no adverse event associated with the use of synbiotics in breast cancer patients during the treatment period(9). Beneficial effects on chemotherapy-induced fatigue and abnormal stool consistency were also observed in subjects receiving synbiotics(9).

Biotin is a water-soluble vitamin that is naturally present in some food and available as a dietary supplement for healthy hair and nails due to its role in keratin production. Most healthy individuals achieve adequate intake of biotin through a well-balanced diet. Current recommendation for biotin by the Food and Nutrition Board (FNB) at the National Academies of Sciences, Engineering, and Medicine stated that the daily adequate intake (AI) for adults is 30 mcg/day. Although biotin has been widely used as dietary supplement, data on the actual benefit of its effect on hair growth is limited(10).

The use of B. longum HK003 in alleviating chemotherapy-induced alopecia in breast cancer patients has not been explored. This pilot, double-blind, randomised, placebo-controlled trial aims to explore on the efficacy and safety of a synbiotic formula (BLHK03) in alleviating chemotherapy-induced alopecia (CIA) in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Females aged between 18 and 60 years who are newly diagnosed with stage I, II or III breast cancer
* Planned chemotherapy including an anthracycline or taxane to be completed within 6 months
* Mentally capable to participate in the study and provide informed consent

Exclusion Criteria:

* Pre-existing female-pattern baldness resembling picture I-3 or higher on the Savin scale at baseline
* History of hair transplantation, psoriasis or severe scalp infection
* Undergoing or plan to receive scalp cooling
* Plan for immunotherapy
* Known pregnancy or lactating
* Severe cardiac, hepatic, renal, pulmonary and haematic lesions or other life-threatening conditions
* Use of antibiotics, probiotics or prebiotics one month prior to enrolment
* No other alternative or complementary treatment for the cancer condition that may affect the gut microbiome analysis
* History of allergy to probiotics or lactose
* History of chemotherapy for other conditions

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-08-18 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with a score of ≤ 2 on the Dean scale (corresponding to hair loss ≤ 50%) 2 months after the final dose of chemotherapy | Baseline to 2 months after the final dose of chemotherapy
  The change of Dean scale (corresponding to hair loss) after chemotherapy compared to baseline. Score 0 means no hair loss and score 4 means all hair is fallen down.

SECONDARY OUTCOMES:
Gut microbial change at 2 months after the final dose of chemotherapy | Baseline to 2 months after the final dose of chemotherapy
  The change of gut microbiota composition at 2 months after the final dose of chemotherapy compared to baseline
Adverse event rates related to the study during the study period | Baseline to 2 months after the final dose of chemotherapy
  The adverse events reported throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Ching, PhD, Study Director — GenieBiome Limited
Locations (2):
- Hong Kong (2):
  - GenieBiome Limited, Hong Kong
  - Heal Medical, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lam S, Zhang J, Yang K, Chu LC, Zhu W, Tang W, Chan FKL, Chan PKS, Wu WKK, Ng SC. Modulation of gut microbiota impacts diet-induced and drug-induced alopecia in mice. Gut. 2022 Nov;71(11):2366-2369. doi: 10.1136/gutjnl-2021-326320. Epub 2022 Jan 5. No abstract available. PMID 34987064
- [Background] Khazaei Y, Basi A, Fernandez ML, Foudazi H, Bagherzadeh R, Shidfar F. The effects of synbiotics supplementation on reducing chemotherapy-induced side effects in women with breast cancer: a randomized placebo-controlled double-blind clinical trial. BMC Complement Med Ther. 2023 Sep 26;23(1):339. doi: 10.1186/s12906-023-04165-8. PMID 37752516
- [Background] Patel DP, Swink SM, Castelo-Soccio L. A Review of the Use of Biotin for Hair Loss. Skin Appendage Disord. 2017 Aug;3(3):166-169. doi: 10.1159/000462981. Epub 2017 Apr 27. PMID 28879195